CLINICAL TRIAL: NCT07028541
Title: To Evaluate the Feasibility of the Clinical Application of Mg-based RemeOs™ DrillPin for Fixation of Fractures of the Distal Radius in Children From the Age of Over 5 and Under 14.
Brief Title: RemeOs™ DrillPin for Fixation of Distal Radius Fractures in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bioretec Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 243-03-CI-02
Record Dates: First submitted 2025-05-22; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Fracture Fixation, Internal; Distal Radius Fracture
Keywords: Distal radius; fracture; RemeOs; DrillPin; Biodegradable Implant
MeSH Terms: conditions — Wrist Fractures; Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Single-arm interventional study in which all enrolled participants receive the investigational device, the RemeOs™ DrillPin, for surgical fixation of distal radius fractures. All patients are followed using a standardized clinical and radiographic assessment schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RemeOs™ DrillPin for Fixation of Distal Radius Fractures (Experimental)
  Interventions: Device: Magnesium-based bioresorbable DrillPin for fixation of distal radius fractures in children

INTERVENTIONS:
Device: Magnesium-based bioresorbable DrillPin for fixation of distal radius fractures in children — This is a first-in-child clinical investigation of a bioresorbable magnesium alloy DrillPin (RemeOs™) for fixation of distal radius fractures in children aged 5 to <14 years. The implant is investigational, not CE-marked or FDA-approved, and represents a novel alternative to traditional metallic implants. It gradually degrades in vivo, eliminating the need for removal. The study focuses on safety and feasibility in a pediatric population, supported by preclinical data from a similar Mg-based RemeOs™ Screw. The DrillPin's material and design are intended to support bone healing without growth disturbances, offering a state-of-the-art, bioresorbable solution tailored for growing patients.

SUMMARY:
This is a pre-market, single-arm, open-label, monocenter clinical investigation evaluating the safety and performance of the magnesium (Mg)-based bioresorbable RemeOs™ DrillPin for surgical fixation of distal radius fractures in pediatric patients. The study will enroll 20 children aged over 5 and under 14 years to assess implantation success, early safety outcomes, and long-term effects on growth and bone healing.

DETAILED DESCRIPTION:
This single-arm, open-label, monocenter clinical investigation is conducted in accordance with ISO 14155 to evaluate the safety and performance of the RemeOs™ DrillPin (a bioresorbable magnesium-based implant) used for internal fixation of distal radius fractures in pediatric patients.

Eligible participants are children aged over 5 and under 14 years who require surgical fixation of a distal radius fracture. The RemeOs™ DrillPin is designed to offer stable fracture fixation while gradually resorbing in the body, potentially reducing the need for implant removal.

Primary objectives include evaluating implantation success-defined by low pain levels (FACES® Pain Rating Scale score <3) and radiographic fracture healing in at least three cortices out of four across two imaging planes at 12 weeks postoperatively-and assessing short-term safety by monitoring adverse events, including device-related and serious adverse events.

Secondary assessments focus on postoperative clinical function and wrist range of motion (ROM), measured using a goniometer, as well as radiographic markers of implant biodegradation. Long-term safety is evaluated through the monitoring of potential growth disturbances at 52 and 104 weeks, including limb length discrepancies or growth plate abnormalities.

This early-stage investigation aims to generate clinical data on the application of magnesium-based resorbable implants in pediatric fracture care and to assess their potential to support bone healing without interfering with skeletal development.

ELIGIBILITY:
Inclusion Criteria:

* Distal Radius Fractures
* Written informed consent of the parent, oral agreement of the patient documented as informant consent of the child
* Subject and parents have been informed of the nature of the study, agrees to participate and parent signs the approved consent form. • Female patients in childbearing age (female patients who have begun menstruation) perform a pregnancy test prior inclusion

Exclusion Criteria:

* Pathological bone lesions (e.g. bone cyst or osteomyelitis)
* Underlying diseases (kidney diseases, uncontrolled diabetes mellitus)
* Polytraumatized patients
* Suspicion of child abuse
* Inability or unwillingness to give informed consent
* Multiple fracture (excluding associated ulna fracture)
* Open Fracture
* Pregnancy (tested in all female patients who have begun menstruation)

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with pain score <3 on the FACES® Pain Rating Scale (criterion of successful implantation) | At 12 weeks postoperatively
  This outcome is one of two predefined criteria used to determine successful implantation. Pain will be measured using the FACES® Pain Rating Scale. A score of less than 3 at 12 weeks postoperatively is considered a successful pain outcome. The FACES® Pain Rating Scale ranges from 0 (no pain) to 10 (worst pain).
Number of participants with radiographic healing in at least 3 of 4 cortices on two-plane radiographs (criterion of successful implantation) | At 12 weeks postoperatively
  This outcome is one of two predefined criteria used to determine successful implantation. Radiographic healing will be assessed at 12 weeks postoperatively using standard anteroposterior and lateral radiographs. Healing is defined as the presence of visible callus formation in at least 3 of the 4 cortices (outer bone surfaces visible on two-plane imaging). Callus formation indicates new bone growth bridging the fracture site, and ≥3 healed cortices reflects adequate fracture consolidation.
Number of participants with at least one adverse event (AE), adverse device effect (ADE), serious adverse event (SAE), or serious adverse device effect (SADE) | From day of surgery through 12 weeks postoperatively
  Safety will be assessed by documenting the occurrence, type, severity, and investigator-assessed relationship to the investigational device or implantation procedure for all adverse events. Events include adverse events (AEs), adverse device effects (ADEs), serious adverse events (SAEs), and serious adverse device effects (SADEs). The assessment will cover the period from surgery through 12 weeks postoperatively and will be based on clinical observations, subject reports, and medical record review.

SECONDARY OUTCOMES:
Passive wrist range of motion (ROM) in degrees measured to assess functional recovery | 2, 4, 6 (optional), 12, 26, 52, and 104 weeks postoperatively
  Passive wrist range of motion (ROM) will be measured in degrees (°) using a goniometer at 2, 4, 6 (optional), 12, 26, 52, and 104 weeks postoperatively. The following directions of movement will be assessed independently: Extension/Flexion, Abduction/Adduction, Pronation/Supination.
  Measurements are recorded separately for the affected wrist and the contralateral (uninjured) wrist. Each direction will be expressed in degrees, and data will be used to evaluate functional recovery of wrist mobility over time.
Number of participants with radiographic evidence of growth disturbance (growth arrest or length discrepancy) | At 52 and/or 104 weeks postoperatively
  Radiographic evaluation for growth disturbance will be performed at 52 and/or 104 weeks postoperatively if clinical assessment suggests axis deviation or deformity. A participant will be recorded as having a growth disturbance if either of the following is observed: Growth arrest or length discrepancy .
  This outcome will be reported as a binary (Yes/No) result per participant.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study data are pseudonymized and retained only by the investigator site with no access to direct identifiers by the sponsor. The sponsor only receives pseudonymized data for analysis and regulatory use.

REFERENCES:
- [Result] Grun NG, Holweg PL, Donohue N, Klestil T, Weinberg AM. Resorbable implants in pediatric fracture treatment. Innov Surg Sci. 2018 May 29;3(2):119-125. doi: 10.1515/iss-2018-0006. eCollection 2018 Jun. PMID 31579775
- [Result] Sturznickel J, Delsmann MM, Jungesblut OD, Stucker R, Knorr C, Rolvien T, Kertai M, Rupprecht M. Safety and performance of biodegradable magnesium-based implants in children and adolescents. Injury. 2021 Aug;52(8):2265-2271. doi: 10.1016/j.injury.2021.03.037. Epub 2021 Mar 18. PMID 33775413
- [Result] Ramoutar DN, Shivji FS, Rodrigues JN, Hunter JB. The outcomes of displaced paediatric distal radius fractures treated with percutaneous Kirschner wire fixation: a review of 248 cases. Eur J Orthop Surg Traumatol. 2015 Apr;25(3):471-6. doi: 10.1007/s00590-014-1553-6. Epub 2014 Oct 21. PMID 25331168
- [Result] Holweg P, Berger L, Cihova M, Donohue N, Clement B, Schwarze U, Sommer NG, Hohenberger G, van den Beucken JJJP, Seibert F, Leithner A, Loffler JF, Weinberg AM. A lean magnesium-zinc-calcium alloy ZX00 used for bone fracture stabilization in a large growing-animal model. Acta Biomater. 2020 Sep 1;113:646-659. doi: 10.1016/j.actbio.2020.06.013. Epub 2020 Jun 14. PMID 32553919